CLINICAL TRIAL: NCT02273375
Title: A Phase III Prospective Double Blind Placebo Controlled Randomized Study of Adjuvant MEDI4736 In Completely Resected Non-Small Cell Lung Cancer
Brief Title: Double Blind Placebo Controlled Controlled Study of Adjuvant MEDI4736 In Completely Resected NSCLC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Intergroupe Francophone de Cancerologie Thoracique (Other); Thoracic Oncology Group of Australasia (TOGA) (Unknown); National Health and Medical Research Council, Australia (Other); National Cancer Institute (NCI), Naples (Unknown); Central and Eastern European Oncology Group (Other); Dutch Society of Physicians for Pulmonology and Tuberculosis (Other); Korean Cancer Study Group (Other); Fundación GECP (Other); West Japan Oncology Group (WJOG) (Unknown); Chinese Thoracic Oncology Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR31; IFCT1401 (Other: Intergroupe Francophone de Cancerologie Thoracique (IFCT)); ACTRN12615000323527 (Registry Identifier: Australian New Zealand Clinical Trials Registry); U1111-1238-5923 (Other: WHO)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI4736 (Experimental): MEDI4736 by intravenous infusion. Treatment from Day 1 for a maximum of 12 months or study drug withdrawal if this occurs earlier.
  Interventions: Drug: MEDI4736
- Placebo (Placebo Comparator): PLACEBO by intravenous infusion. Treatment from Day 1 for a maximum of 12 months or study drug withdrawal if this occurs earlier
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI4736
  Arms: MEDI4736
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out whether it is better to receive a new drug, MEDI4736, or better to receive no further treatment after surgery (and possibly chemotherapy) for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of primary non-small cell carcinoma of the lung. according to WHO Classification of Tumours (WHO Classification of Tumours of the Lung, Pleura, Thymus and Heart. WHO/IARC Classification of Tumours, 4th Edition, Volume 7). Patients with large-cell neuroendocrine carcinomas are not eligible.
* Patients must be classified post-operatively as Stage IB (≥ 4cm in the longest diameter), II or IIIA on the basis of pathologic criteria. Note: Although T3N2M0 tumours have been reclassified to stage IIIB in the 8th edition of the IASLC staging system, these patients remain eligible (as stage IIIA under the 7th edition criteria).

  * Complete surgical resection of the primary NSCLC is also mandatory. All gross disease must have been removed at the end of surgery. All surgical margins of resection must be negative for tumour. Resection may be accomplished by open or VATS techniques

Note: Patients with synchronous primary tumours will not be eligible due to the potential uncertainty regarding their appropriate PD-L1 status.

Prior Systemic Therapy:

* Pre-operative (neo-adjuvant) platinum based or other chemotherapy is not permissible.
* Patients may have received prior post-operative platinum based chemotherapy as per standard of care.
* No prior anticancer therapy for treatment of NSCLC other than standard post-operative adjuvant chemotherapy is permissible.

Radiation:

• Patients with N2 disease only who receive adjuvant post-operative radiation therapy are eligible provided they meet the protocol specified timing criteria for surgery, adjuvant chemotherapy and randomization. Pre-operative radiation therapy is not permissible.

* The patient must have an ECOG performance status of 0, 1.
* Hematology: . Absolute neutrophil count ≥ 1.5 x 109/L or ≥ 1,500/µl Platelets ≥ 100 x 109/L or ≥ 100,000/µl
* Biochemistry:

Total bilirubin* ≤ institutional upper limit of normal Alkaline phosphatase ≤ 2.5 x institutional upper limit of normal AST(SGOT) and ALT(SGPT) ≤ 2.5 x institutional upper limit of normal Creatinine Clearance ≥ 40 ml/min

* excluding Gilbert's syndrome

Creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by Cockcroft Formula:

Females: GFR = 1.04 x (140-age) x weight in kg serum creatinine in μmol/L Males: GFR = 1.23 x (140-age) x weight in kg serum creatinine in μmol/L

* Patient able and willing to complete the QoL, economics and other questionnaires. The baseline assessment must already have been completed within required timelines prior to randomization. Inability (illiteracy, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Patients must be accessible for treatment and follow-up. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, adverse events, and follow-up
* Protocol treatment is to begin within 2 working days of patient randomization

Exclusion Criteria:

* Patients with a history of other malignancies, except:

  * adequately treated non-melanoma skin cancer,
  * curatively treated in-situ cancer, or
  * other malignancies curatively treated with no evidence of disease for ≥ 5 years following the end of treatment and which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
* A combination of small cell and non-small cell lung cancer, pulmonary carcinoid tumour or large-cell neuroendocrine carcinoma (LCNEC).
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. NOTE: patients with Grave's disease and/or psoriasis not requiring systemic therapy within the last two years from randomization and patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement are not excluded.
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of randomization* or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy.
* Live attenuated vaccination administered within 30 days prior to randomization.
* History of hypersensitivity to MEDI4736 or any excipient.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction within the previous year or cardiac ventricular arrhythmias requiring medication, history of 2nd or 3rd degree atrioventricular conduction defects). Patients with a significant cardiac history, even if controlled, must have a LVEF > 50% within 12 weeks prior to randomization.
* Concurrent treatment with other investigational drugs or anti-cancer therapy.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol. This includes but is not limited to:

  * known clinical diagnosis of tuberculosis;
  * known active hepatitis B infection (positive HBV surface antigen (HBsAg)). Patients with a past or resolved hepatitis B infection (defined as presence of hepatitis B core antibody (anti-HBc) and absence of HBSAg) are eligible;
  * known active hepatitis C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA;
  * known human immunodeficiency virus infection (positive HIV antibodies).
  * known pneumonitis or pulmonary fibrosis with clinically significant impairment of pulmonary function
* Pregnant or lactating women. Women of childbearing potential must have a urine pregnancy test proven negative within 14 days prior to randomization. Men and women of child-bearing potential must agree to use adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1415 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Compare Disease free survival (DFS) for patients with NSCLC that is PD-L1 expression TC ≥ 25% and patients without common activating EGFR mutations or ALK gene rearrangements | 6.7 years

SECONDARY OUTCOMES:
Disease-free survival in the remaining 5 patient sub-populations defined by PD-L1 expression levels and EGFR/ALK status | 8 years
  (PD-L1 TC ≥ 1% and patients without common activating EGFR mutations or ALK gene rearrangements; all patients without common activating EGFR mutations or ALK gene rearrangements; all PD-L1 TC ≥ 25%; all PD-L1 TC ≥ 1%; all randomized patients)
Compare overall survival (OS) for patients in the six patient sub-populations defined by PD-L1 expression levels and EGFR/ALK status | 8 years
Compare Lung cancer specific survival for patients in the six patient sub-populations defined by PD-L1 expression levels and EGFR/ALK status | 8 years
Evaluate the nature, severity and frequency of adverse effects and tolerability of MEDI4736 | every 6 months
  All patients who receive at least one dose of MEDI4376/placebo will be included in the safety analysis. Descriptive summary tables will be presented on safety parameters by treatment arm. There will be safety monitoring by the CCTG Data Safety Monitoring Committee (DSMC) every 6 months
Evaluate the Quality of life in the six patient sub-populations defined by PD-L1 expression levels and EGFR/ALK status | 8 years
  The quality of life (QoL) of patients will be assessed using EORTC QLQ-C30 and the lung cancer module (QLQ-LC13) incorporated.
Determine survival benefits participants judge necessary to make adjuvant immunotherapy worthwhile | 8 years
Determine the incremental cost effectiveness and cost utility ratios for MEDI4736 | 8 years
Evaluate the predictive/prognostic significance of PD-L1 expression | 8 years
Evaluation of changes in plasma/serum cytokines and other blood and tissue based biomarkers after treatment with MEDI4736 and at disease event | 8 years
Explore polymorphisms that may be associated with outcomes | Baseline only

CONTACTS AND LOCATIONS:
Overall Officials: Glenwood Goss, Study Chair — Ottawa Hospital Research Institute, Ontario, Canada
Locations (271):
- United States (9):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - USC Norris/Comprehensive Cancer Centre, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Duke University Medical Center, Durham, North Carolina
  - Hematology and Oncology Associates of NEPA, Dunmore, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Reading Hospital Medical Center, West Reading, Pennsylvania
- Australia (27):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Coffs Habour Health Campus - NCCI, Coffs Harbour, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St. George Hospital, Cancer Care Centre, Kogarah, New South Wales
  - Liverpool Cancer Therapy Centre, Liverpool Hospital, Liverpool, New South Wales
  - Northern Cancer Institute St Leonards, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Mater Medical Centre, Brisbane, South, QLD
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - Frankston Hospital - Peninsula Oncology Centre, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital Research Foundation, Parkville, Victoria
  - Epworth HealthCare - Richmond, Richmond, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - St John of God Subiaco, Subiaco, Western Australia
  - Flinders Medical Center, Adelaide
  - Canberra Hospital, Garran
  - St. Vincent's Hospital, Victoria Park
- Brazil (10):
  - Suporte Nutricional e Quimioterapia LTDA PRONUTRIR, Fortaleza, Ceará
  - Hospital Evangelico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Cetus Hospital Dia Oncologia, Belo Horizonte, Minas Gerais
  - Liga Norte Riograndense Contra o Cancer, Natal, Rio Grande do Norte
  - Instituto Tacchini de Pesquisa em Saude, Bento Gonçalves, Rio Grande do Sul
  - Centro de Oncologia e Radioterapia (COR) Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Faculdade de Medicina do ABC, São Paulo, Santo Andre
  - Fundacao Faculdade Regional de Medicina, São José do Rio Preto, São Paulo
  - Instituto Nacional de Cancer (INCA), Rio de Janeiro
- Bulgaria (3):
  - MHAT Serdika - Medical Oncology Clinic, Sofia
  - MHAT Nadezhda Hospital, Sofia
  - Medical Centre Synexus, Sofia
- Canada (33):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Sciences Centre/Thunder, Thunder Bay, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - PEI Cancer Treatment Centre, Charlottetown, Prince Edward Island
  - Lévis, Quebec
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - Centre Integre Universitaire De Sante Et De Services, Montreal, Quebec
  - University Institute of Cardiology and, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- China (17):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Province Cancer Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hosp of Shantou Medical Colleg, Shantou, Guangdong
  - The People Hospital of Guangxi Zhuang Autonomous Reg, Nanning, Guangxi
  - Henan province Cancer Hospital, Zhengzhou, Henan
  - The Second Xiangya Hospital of Central South Univer, Changsha, Hunan
  - The First People Hospital of Yueyang, Yueyang, Hunan
  - Nanjing General Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital Of Xuzhou Medical College, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu People Hospital, Yangzhou, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital Of Qingdao University, Qingdao, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Yunnan Provincial Cancer Hospital, Kunming, Yunnan
  - Sir run run shaw hospital School of Medicine, Hangzhou, Zhejiang
- France (54):
  - CRLCC - Paoli-Calmette, Marseille, BP
  - Hopital de la Croix-Rousse, Lyon, Cedex 04
  - Centre hospitalier universitaire de Montpellier, Montpellier, Cedex 05
  - AP-HP Hopital Tenon, Paris, Cedex 20
  - Hopital Albert Michallon, Grenoble, Cedex 9
  - CHRU de Tours - Hopital Bretonneau, Tours, Tours Cedex 9
  - CHU - Angers, Angers
  - Centre Hospitalier - Avignon, Avignon
  - Institut Sainte Catherine, Avignon
  - Bayonne - Centre Hospitalier, Bayonne
  - Hopital Jean Minjoz, Besançon
  - Hopital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord, Bordeaux
  - Boulogne - Ambroise Pare, Boulogne
  - Caen - CHU, Caen
  - Centre Hospitalier de Chambery, Chambéry
  - Centre Hospitalier de Cholet, Cholet
  - HIA Percy, Clamart
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - Hopital Louis Pasteur, Colmar
  - Annemasse - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - CHU Hopital du Bocage, Dijon
  - Centre Hospitalier Intercommunal - Elbeuf, Elbeuf
  - Centre Hospitalier departemental, La Roche-sur-Yon
  - Versailles - CH Andre Mignot, Le Chesnay
  - Centre Hospitalier du Mans, Le Mans
  - Lille - Hopital Calmette, Lille
  - Centre Hospitalier Lyon Sud, Lyon
  - Hopital Europeen, Marseille
  - Marseille - Hopital Nord, Marseille
  - Centre Hospitalier les Chanaux, Mâcon
  - CH de la Region d'Annecy, Metz-Tessy
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Centre Antoine Lacassagne - Nice, Nice
  - Centre Hospitalier Regional Hopital de la Source, Orléans
  - Hopital Saint Louis, Paris
  - Fondation Hopital Saint Joseph, Paris
  - Paris - HEGP, Paris
  - Paris - Institut Curie, Paris
  - Hopital Bichat, Paris
  - Centre Hospitalier General de Pau, Pau
  - Centre Hospitalier de Perigueux, Périgueux
  - Centre Hospitalier Rene Dubos, Pontoise
  - CHU de Rouen, Rouen
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Nouvel Hopital Civil Hopitaux, Strasbourg
  - Suresnes - Foch, Suresnes
  - Thonon-les-Bains - Hopital Georges Pianta, Thonon-les-Bains
  - CHITS Toulon Sainte Musse, Toulon
  - Hopital Larrey, Toulouse
  - Villefranche sur Saone - CH, Villefranche-sur-Saône
- Semmelweis University Pulmonology Department, Budapest, Hungary
- Italy (27):
  - AOU Ospedali Riuniti Umberto I, Torrette, AN
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino, AV
  - IRCCS Ospedale Oncologico Giovanni Paolo II, Bari, BA
  - Instituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Ospedale S. Paolo - U.O. di Oncologia Medica, Milan, MI
  - Azienda Ospedaliera di Perugia Santa Maria, Perugia, PG
  - Centro di Riferimento Oncologico - CRO, Aviano, PN
  - Fondazione Salvatore Maugeri Oncologia Medica, Pavia, PV
  - OUC Oncologia Medica - Presidio Ospedaliero, Ravenna, RA
  - Oncologia Medica IRCCS Arcispedale Maria, Reggio Emilia, RE
  - Istituti Fisioterapici Ospitalieri IFO Istituto, Rome, RM
  - A.O. Busto Arsizio - P.O. Saronno, Saronno, VA
  - AOU Integrata Verona Policlinico GB, Verona, VR
  - U.O. di Oncologia Medica Azienda Ospedaliera G Rummo, Benevento
  - PO A Perrino ASL Brindisi - UOC Oncologia Medica, Brindisi
  - AOU Policlinico Vittorio Emanuele UOC di Oncologia, Catania
  - U.O. di Oncologia Ospedale Villa Scassi, Genova
  - Intstituto Scientifico Romangnolo, Meldola
  - European Institute of Oncology, Milan
  - U.O.C. di Oncologia U.L.S.S. 13, Mirano
  - Azienda Ospedaliera di Rilievo Nazionale, Napoli
  - Dott. Fortunato Ciardiello,Cattedra Oncologia Medica, Napoli
  - Unita Sperimentazioni Cliniche Istituto per lo, Napoli
  - Universita Federico II UOC Oncologia Medica, Napoli
  - UOC Oncologia Medica II Instituto Oncologio Veneto, Padua
  - Azienda USL di Piacenza, Ospedale Gugliemimo Salieto, Piacenza
  - Azienda Ospedaliera S. Camillo-Forlanin, Rome
- Japan (28):
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Hospital of the University of Occupational and, Kitakyushu, Fukuoka
  - Gifu Univiesity Hospital, Gifu, Gifu
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Kure Medical Center, Kure, Hiroshima
  - Koube University Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine, Nishinomiya-shi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kinki University Hospital Faculty of Medicine, Ōsaka-sayama, Osaka
  - National Hospital Organization Kinki-Chuo, Sakai, Osaka
  - Tottori University Hospital, Yonago, Tottori
  - National Hospital Organization Yamaguchi, Ube, Yamaguchi
  - Chiba University Hospital, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Osaka City General Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Juntendo University Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Netherlands (9):
  - Universitair medisch centrum Nijmegen st Radboud, Nijmegen, Gelderland
  - Amphia ziekenhuis, Breda, North Brabant
  - Tergooi locatie Hilversum, Hilversum, North Holland
  - Isala, Zwolle, Overijssel
  - Netherlands Cancer Institute, Amsterdam
  - Free University Hospital, Amsterdam
  - UMC Groningen, Groningen
  - Academical Hospital Maastricht, Maastricht
  - Erasmus Medical Center (EMC), Rotterdam
- Christchurch Hospital, Christchurch, New Zealand
- Poland (3):
  - Klinika Onkologii i Radioterapii Uniwersyteckie, Gdansk
  - Specjalistyczny Szpital im, Szczecin
  - Samodzielny Publiczny Szpital Specjalistyczny, Zakopane
- Romania (8):
  - Conformal Med Terra HIFU, Bucharest
  - Spitalul de Psihiatrie Dr. Constantin Gorgos, Bucharest
  - Oncology Institute Bucharest, Bucharest
  - Oncological Institute "Ion Chiricuta", Cluj-Napoca
  - OCH - Ovidius Clinical Hospital, Constanța
  - Centrul de Oncologie Sf Nectarie, Craiova
  - SC Oncolab SRL, Craiova
  - Spital Lotus SRL, Ploieşti
- National University Hospital, Singapore, Singapore
- South Korea (9):
  - Keimyung University Dongsan Medical Center, Daegu, Dalseogu
  - Chung Ang University Hospital, Seoul, Dongjak Gu
  - Veterans Health Service Medical Center, Seoul, Gangdong-gu
  - The Catholic University of Korea Bucheon, Bucheon-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Uijeongbu ST Marys Hospital, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul
  - The Catholic University of Korea,, Seoul
- Spain (17):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Insular de Gran Canaria, Las Palmas, Gran Canaria
  - Hospital Teresa Herrera, A Coruña
  - Hospital General de Alicante, Alicante
  - Hoapital Quiron Dexeus, Barcelona
  - Hospital Vall d Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Universitario la Princesa, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital General Universitario de Valencia, Valencia
- Taiwan (11):
  - Far Eastern Memorial Hospital, New Taipei City;, Taiwan
  - Chang-Gung Memorial Hospital - Chiayi, Chiayi City
  - Kaohsiung Medical University, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Chang-Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Mackay Memorial Hospital, Taipei
  - Veterans General Hospital - Taipei, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang-Gung Memorial Hospital - Linkou, Taoyuan District
- Ukraine (3):
  - Dnipropetrovsk City Clinical Hospital No.4, Dnipropetrovsk
  - Regional Oncology Center, Sumy
  - Vinnytsia Regional Clinical Oncology Dispensary, Vinnitsia

IPD SHARING:
Plan to Share IPD: No